CLINICAL TRIAL: NCT04413747
Title: Yoga- Based Breathing for Vagus Nerve Stimulation as Home-care Adjuvant Treatment Against Burden COVID-19
Brief Title: Yoga Pranayama Adjuvant to Treat Burden COVID-19
Acronym: YOCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Health Ricerca e Sviluppo S.R.L. (Industry)
Collaborators: Swami Vivekananda Yoga Anusandhana Samsthana, Bangaluru , India (Unknown); Yoga Experience Association,Cervia (Ra), Italy (Unknown); EJTN GEIE, Brussellese, Belgium (Unknown); Casa di Riposo e Ambulatorio Giardino St Lucia, Massa Lomabarda (Ra) Italy (Unknown); Halnet Srl, Faenza (Ra), Italy (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020_COVID-19_YOGA
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Coronavirus Infection; Cytokine Storm; Mental Disorder
Keywords: COVID-19; CYTOKINE STORM; MEDICAL YOGA PRANAYAMA; VAGUS NERVE STIMOLATION; MENTAL DISORDER
MeSH Terms: conditions — Coronavirus Infections; Cytokine Release Syndrome; Mental Disorders; COVID-19

STUDY DESIGN:
Intervention Model Description: Prospective cohort study based on clinical assessment. Model- based adjusted outcome via hierarchical comparison of control curves using COVID19 national epidemic data with cyber layer algorithm of population
Masking Description: identifier number (ID) without any refer to clinical assessment or to patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga-based breathing support (Experimental): Three daily yoga pranayama breathing cycles within existing home-care provision of Covid19's patients (protocols shared dated 27 March 2020 by Italian Society of Infectious and Tropical Diseases - Italian General Practitioners Physician - Italian Society of General Medicine, Italy)
  Interventions: Behavioral: morning Yoga-based breathing support; Behavioral: pre_lunch Yoga-based breathing support; Behavioral: pre_dinner Yoga-based breathing support

INTERVENTIONS:
Behavioral: morning Yoga-based breathing support — Low and deep inspiration and phonetic syllable OM laryngeal vibration ( OM technique) as expiratory exercises, sitting in easy pose. The length of more than 5 -8 sec. and frequency between 20 and 23 breaths /min. Conscious breath number (n°) of 15 respiratory acts (RAc) and OM technique n° of 5 RAc and Bhramari pranayama n° of 5 RAc.
  Other Names: First procedure
Behavioral: pre_lunch Yoga-based breathing support — Low and deep inspiration and OM technique as expiratory exercises, sitting in easy pose.The length of more than 5 -8 sec. and frequency between 20 and 23 breaths /min. Conscious breath number (n°) of 15 respiratory acts (RAc) and OM technique n° of 5 RAc and Surya Bheda pranayama n° of 5 RAc.
  Other Names: Second procedure
Behavioral: pre_dinner Yoga-based breathing support — Low and deep inspiration and OM technique as expiratory exercises, sitting in easy pose.The length of more than 5 -8 sec. and frequency between 20 and 23 breaths /min. Conscious breath number (n°) of 15 respiratory acts (RAc) and OM technique n° of 5 RAc and Nadi Shodhana pranayama n° of 5 RAc.
  Other Names: Third procedure

SUMMARY:
COronaVIrus Disease or Severe Acute Respiratory Syndrome -CoV-2 or COVID-19, mortality occurs mainly from immunological behavior or by suicide after healing . In both cases, the causal link is coronavirus within the host response. The rationale of use of deep yoga breathing as adjuvant treatment to COVID-19 disease , is linked to the mechanical action to stimulate the vagus nerve through scalene and sternocleidomastoid muscles function of which the continuity of action bring to modulate upto suppress, the inflammatory reflex and pro-inflammatory cytokines overproduction and contextual lowering of the sympathetic stress response as a first cause of sleep and late mental disorders which can increase the annual suicide rate. An easily breathing medical Yoga protocol has been developed to test a cost-effective care provision, training, contact tracing and mass efficacy testing.

DETAILED DESCRIPTION:
COronaVIrus Disease or Severe Acute Respiratory Syndrome -CoV-2 or COVID-19, pandemic threatens patients, societies and healthcare systems around the world. Morbidity and lethality have a direct link with the early vicious circles triggered by an acute microcirculation endotheliopathy, a correlated coagulopathy, up to late hypoxic damage of multi organ tissue The host immunity determines the progress of the disease , its lethality and the need of care intensity. The clinical course of the infection consist of three stage of which only the third -which intervenes in a low incidence of patients - need of hospitalization for severe hyperinflammatory syndrome including acute respiratory failure, while first and the second or moderate pulmonary involvement, might manage and monitoring within a homecare program during quarantine. Actually, the rough mortality in Italy is - at the current date - 7.6 % with an expected death of 0.004 of the whole population. The late lethality - still little known - from COVID-19 is to be correlated with mental disorders from stress response emerging from the first three COVID-19's stages and which result in a significant increase in suicides that is estimated at 30% more than expected of 7.4 deaths for 100,000 residents. This estimate can be considered as stage 4 of the disease or post COVID-19 mortality. In this scenario, mortality of COVID-19 is by intensity response of "the host " and in the meantime, a cutoff for homecare, hospitalization and time-related stress disease. Lines of evidence reports that direct-indirect stimulation of vagus nerve bring to the modulating of pro-inflammatory cytokines with effective systemic anti-inflammatory effect and has shown antidepressant effects in chronic treatment resistant depression. Because the vagus nerve is linked to brain regions important in anxiety regulation (locus coeruleus, orbitofrontal cortex, insula, hippocampus and amygdala), this pathway is involved in perceiving various somatic and cognitive symptoms that characterize anxiety and mental disorder disorders. On the basis of all these reasoning we plan to introduce a medical based-yoga deep breathing for activation of vagus nerve by scalene and sternocleidomastoid muscles function during breathing, as an adjuvant of care of the 1-2 and 4 stages of the COVID-19 disease to counteract the cumulative incidence of mortality and better outcome. Medical yoga protocol has been developed and designed to test a cost-effective care provision, training, contact tracing and mass efficacy testing.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial;
* Male or Female, aged 18 years or above;
* Diagnosed COVID-19's infection;
* Informed consent;
* Having been diagnosed in the last 1 week;
* In the Investigator's opinion, is able and willing to comply with all trial requirements;
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the trial;
* Patients who continue to be followed at home.

Exclusion Criteria:

The participant may not enter the trial if ANY of the following apply:

* No informed consent;
* Participant is not willing and able to give informed consent for participation in the trial;
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial;
* Hospitalization patients;
* Having a serious cognitive impairment;
* Having serious hearing and vision problems;
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial;
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-08-15 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | 12 months.
  COVID-19's Patients mortality all cause: incidence proportion.
Mortality-suicide | 12 months.
  COVID-19's Patients suicide: incidence proportion.

SECONDARY OUTCOMES:
Incidence of hospitalization for respiratory failure of COVID-19's Patients- | 1 months.
  In-hospital COVID-19's Patients oxygen invasive ventilation or high flow oxygen devices :incidence proportion of Brescia COVID-19 respiratory Severity Scale Index (Levels 0-3 worse outcome) cutoff Level ≥ 2 -
Incidence of al home professional psychiatric-psychological interventions for mental disorder. | 12 months.
  Homecare interventions for anxiety and depression requiring drugs treatment: incidence proportion.
Incidence of mental disorder: Beck Depression Inventory-Second Edition (BDI-II). | 12 months.
  Scoring system for depression and anxiety requiring drugs treatment: incidence proportion of BDI-II aggregate components score 0- 63 ( worse outcome) , cutoff > 29.
Incidence od spleep disorder:Pittsburgh Sleep Quality Index (PSQI). | 12 months.
  Scoring system for sleep disorders requiring drugs treatment: incidence proportion of aggregate PSQI score 0-21 (worse outcome) , cutoff > 8.

CONTACTS AND LOCATIONS:
Overall Officials: Nagarathna Raghuram, MD, Principal Investigator — Vivekananda Yoga Anusandhana Samsthana, Bengaluru, India; HR Nagendra., Eng, Study Chair — Vivekananda Yoga Anusandhana Samsthana, Bengaluru, India; Maria Donatella Barbagallo, MD, Principal Investigator — Yoga Experience Association,Cervia (Ra), Italy; Enrico Ricci, MD, Principal Investigator — Yoga Experience Association,Cervia (Ra), Italy; Morena Gaddoni, MD, Principal Investigator — Casa di Riposo Giardino St Lucia, Massa Lombarda (Ra) Italy; Maria Luisa Vitobello, Study Director — EJTN GEIE, Brussellese, Belgium; Luca Ghetti, Eng., Study Director — Halnet Srl; Fabio Zucchetta, MD, Principal Investigator — Casa di Riposo Giardino St Lucia, Massa Lombarda (Ra) Italy
Locations (1):
- Ambulatorio Telemedicina Giardino St Lucia, Massa Lombarda, Ravenna, Italy

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study will be available upon request within a web_ client structure
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 18 months
Access Criteria: ID (nikname ) and password
URL: https://ifc.cnr.it

REFERENCES:
- [Background] Wenham C, Smith J, Morgan R; Gender and COVID-19 Working Group. COVID-19: the gendered impacts of the outbreak. Lancet. 2020 Mar 14;395(10227):846-848. doi: 10.1016/S0140-6736(20)30526-2. Epub 2020 Mar 6. No abstract available. PMID 32151325
- [Background] Johansson PI, Stensballe J, Ostrowski SR. Shock induced endotheliopathy (SHINE) in acute critical illness - a unifying pathophysiologic mechanism. Crit Care. 2017 Feb 9;21(1):25. doi: 10.1186/s13054-017-1605-5. PMID 28179016
- [Background] Borovikova LV, Ivanova S, Zhang M, Yang H, Botchkina GI, Watkins LR, Wang H, Abumrad N, Eaton JW, Tracey KJ. Vagus nerve stimulation attenuates the systemic inflammatory response to endotoxin. Nature. 2000 May 25;405(6785):458-62. doi: 10.1038/35013070. PMID 10839541
- [Background] Koopman FA, Chavan SS, Miljko S, Grazio S, Sokolovic S, Schuurman PR, Mehta AD, Levine YA, Faltys M, Zitnik R, Tracey KJ, Tak PP. Vagus nerve stimulation inhibits cytokine production and attenuates disease severity in rheumatoid arthritis. Proc Natl Acad Sci U S A. 2016 Jul 19;113(29):8284-9. doi: 10.1073/pnas.1605635113. Epub 2016 Jul 5. PMID 27382171
- [Background] Thayer JF, Sternberg EM. Neural aspects of immunomodulation: focus on the vagus nerve. Brain Behav Immun. 2010 Nov;24(8):1223-8. doi: 10.1016/j.bbi.2010.07.247. Epub 2010 Jul 30. PMID 20674737
- [Background] Lv H, Zhao YH, Chen JG, Wang DY, Chen H. Vagus Nerve Stimulation for Depression: A Systematic Review. Front Psychol. 2019 Jan 31;10:64. doi: 10.3389/fpsyg.2019.00064. eCollection 2019. PMID 30766497
- [Background] O'Reardon JP, Cristancho P, Peshek AD. Vagus Nerve Stimulation (VNS) and Treatment of Depression: To the Brainstem and Beyond. Psychiatry (Edgmont). 2006 May;3(5):54-63. PMID 21103178
- [Background] Jordana J, Trivino-Salazar JC. Where are the ECDC and the EU-wide responses in the COVID-19 pandemic? Lancet. 2020 May 23;395(10237):1611-1612. doi: 10.1016/S0140-6736(20)31132-6. Epub 2020 May 13. No abstract available. PMID 32410757
- [Background] Zhu S, Wu Y, Zhu CY, Hong WC, Yu ZX, Chen ZK, Chen ZL, Jiang DG, Wang YG. The immediate mental health impacts of the COVID-19 pandemic among people with or without quarantine managements. Brain Behav Immun. 2020 Jul;87:56-58. doi: 10.1016/j.bbi.2020.04.045. Epub 2020 Apr 18. PMID 32315758
- Available data/document: Study Protocol: guest_1 — http://giardinostlucia.it
- Available data/document: Informed Consent Form: guest_2 — http://giardinostlucia.it
- Available data/document: Individual Participant Data Set: guest_3 — http://giardinostlucia.it